CLINICAL TRIAL: NCT06262438
Title: A Phase II, Single Arm, Open Label, Study on the Safety, Efficacy, Pharmacokinetics & Pharmacodynamics of Quizartinib + Chemotherapy and as Single-agent After High Dose Therapy in Newly Diagnosed Pediatric FLT3-ITD+ and NPM1wt AML Patients
Brief Title: CHIP-AML22/Quizartinib: Quizartinib + Chemotherapy in Newly Diagnosed Pediatric FLT3-ITD+ and NPM1wt AML Patients
Acronym: CHIP-AML22/Q
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH22CAQ; 2022-002886-14 (EudraCT Number); 2023-505000-27 (Other: EU CT Number)
Record Dates: First submitted 2024-01-26; First posted 2024-02-16 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia in Children
Keywords: FLT3-ITD+ NPM1wt AML
MeSH Terms: interventions — quizartinib; Etoposide; Dexrazoxane; Mitoxantrone; Cytarabine; Methotrexate; Daunorubicin; fludarabine

STUDY DESIGN:
Intervention Model Description: Given the rarity of pediatric subjects with newly diagnosed Acute Myeloid Leukemia (AML) with FLT3-ITD mutations and the slow enrollment in historical studies, it is not feasible to enroll a sufficient number of subjects for an adequately powered randomized study. Therefore, a standard oncology Phase 2 response-rate design has been chosen. One of the exploratory objectives planned is to compare the outcome of patients treated in this study to the outcome of patients treated in the NOPHO-DBH AML-2012 study as historical control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Quizartinib (Experimental): Quizartinib will be administered for 14 days following the completion of standard of care chemotherapy for up to 3-5 cycles of induction and consolidation. After high dose chemotherapy or allo-Stem Cell Transplantation (allo-SCT), patients will receive continuation treatment with quizartinib for six 28-day courses
  Interventions: Drug: Quizartinib; Drug: Etoposide; Drug: Dexrazoxane; Drug: Mitoxantrone; Drug: Cytarabine; Drug: Methotrexate; Drug: Daunorubicin; Drug: Fludarabine; Other: allo-SCT

INTERVENTIONS:
Drug: Quizartinib — Quizartinib is a novel oral Class III receptor tyrosine kinase (RTK) inhibitor exhibiting highly potent and selective but reversible inhibition of FMS-like tyrosine kinase FLT3. The dose will be adjusted for the patient's body weight (BW) as measured at the start of each course. Quizartinib will be administered orally once daily and is taken for 14 consecutive days during induction and consolidation courses.
  Induction course 1: Start on day 13; Induction course 2: Start on day 9; Consolidation course 1: Start on day 6; Consolidation courses 2 and 3 (only if no allo-SCT is done): Start on day 6.
  Continuation courses 1-6: patients will receive quizartinib for six 28-day courses. For the first 15 days of course 1 a starting dose will be applicable. On course 1 Day 16, the dose will be increased if the average QTc of the triplicate Electrocardiograms is ≤450 msec on course 1 Day 15. Once the dose is increased, the patient may continue on this dose as long as dose reduction is not needed.
  Other Names: AC220; Quizartinib dihydrochoride; Vanflyta
Drug: Etoposide — Induction course 1: 150 mg/m2 once daily by Intravenous (IV) infusion over 2 hours (+/- 30 mins) on days 1-5 inclusive (total 5 doses).
  Induction course 2: 150 mg/m2 once daily by IV infusion over 2 hours (+/- 30 mins) on days 6-8 inclusive (total 3 doses).
  Consolidation course 2 (only if no allo-SCT is done): 100 mg/m2 once daily by IV infusion over 1 hour (+/- 15 mins) on days 1-5 inclusive (total 5 doses).
Drug: Dexrazoxane — Induction course 1: 250 mg/m2 once daily by 15 mins IV infusion shortly before Mitoxantrone on day 6-10 inclusive (total 5 days), per investigator discretion and per institutional guidelines and availability.
  Induction course 2: 600 mg/m2 once daily by 15 mins IV infusion shortly before daunorubicin on day 2,4,6 inclusive (total 3 does), per investigator discretion and per institutional guidelines and availability.
  Consolidation course 1: 500 mg/m2 once daily by 15 mins IV infusion shortly before Mitoxantrone on 3-5 inclusive (total 3 does), per investigator discretion and per institutional guidelines and availability.
Drug: Mitoxantrone — Induction course 1: 5 mg/m2 once daily by IV infusion over 1 hour (+/- 15 mins) on days 6-10 inclusive (total 5 doses). Please note that mitoxantrone and cytarabine should not be given concomitantly. Mitoxantrone should be completed before cytarabine is given.
  Consolidation course 1: 10 mg/m2 once daily by IV infusion over 1 hour (+/- 15 mins) on days 3-5 inclusive (total 3 doses).
Drug: Cytarabine — Induction course 1: 200 mg/m2 once daily by IV infusion over 12 hours (+/- 1 hour) on days 6-12 inclusive (total 7 doses), following mitoxantrone. Induction course 2: 100 mg/m2 once daily by continuous IV infusion on days 1-2 inclusive. And 100 mg/m2 twice daily as a 30min (+/- 10 mins) IV infusion every 12 hours on days 3-8 inclusive (total 12 doses). Consolidation course 1: 1000 mg/m2 twice daily by IV infusion over 2 hours (+/- 30 min) every 12 hours on days 1-3 inclusive (total 6 doses).
  Consolidation course 2 (only if no allo-SCT is done): 3000 mg/m2 twice daily by IV infusion over 2 hours (+/- 30 mins) every 12 hours on days 1-3 inclusive (total 6 doses).
  Consolidation course 3 (only if no allo-SCT is done): 2000 mg/m2 once daily by IV infusion over 3 hours (+/- 1 hour) starting 4 hours after fludarabine on days 1-5 inclusive (total 5 doses), following fludarabine.
Drug: Methotrexate — Induction course 1: Methotrexate (MTX) Intrathecal therapy (IT) prophylaxis is age-adjusted. If MTX is given at diagnosis omit IT therapy on day 6 unless in case of CNS involvement (CNS3). For children with initial CNS involvement (CNS3) MTX IT is replaced with triple IT and given more frequently. For children with CNS2, CSF must be investigated on day 22; if leukemic cells persist, treat as CNS3.
  Induction course 2, Day 1: MTX (IT) prophylaxis is age-adjusted. For children with initial CNS involvement (CNS3) MTX IT is replaced with triple IT and given more frequently.
  Consolidation course 1, Day 1: MTX (IT) prophylaxis is age-adjusted. For children with initial CNS involvement (CNS3) MTX IT is replaced with triple IT and given more frequently.
  Consolidation course 2 and 3, Day 1 (only if no allo-SCT is done): MTX (IT) prophylaxis is age-adjusted. For children with initial CNS involvement (CNS3) MTX IT is replaced with triple IT and given more frequently.
Drug: Daunorubicin — Induction course 2: 60 mg/m2 once daily by IV infusion over 1 hour (+/- 15 mins) on days 2,4,6 inclusive (total 3 doses).
Drug: Fludarabine — Consolidation course 3 (only if no allo-SCT is done): 30 mg/m2 once daily by IV infusion over 30 mins (+/- 10 mins) on days 1-5 inclusive (total 5 doses).
Other: allo-SCT — The SCT procedure is left to the discretion of the investigator and not part of this protocol.

SUMMARY:
The CHIP-AML22 Master protocol has the overall aim of increasing the cure rate in newly diagnosed pediatric de novo AML patients, while avoiding unnecessary toxicity. The linked Quizartinib trial (CHIP-AML22/Quizartinib) is a phase II, single arm, open label, study on the safety, efficacy, pharmacokinetics and pharmacodynamics of quizartinib in combination with chemotherapy and as single-agent after high dose therapy in newly diagnosed pediatric AML patients with a FLT3-ITD mutation and NPM1 wild-type.

DETAILED DESCRIPTION:
The CHIP-AML22/Quizartinib study is a single-arm, multinational, multicenter, open-label phase II study, with a safety run-in, aiming to assess the safety, efficacy, pharmacokinetics and pharmacodynamics of quizartinib, a FLT3-inhibitor, as IMP added to standard of care chemotherapy in newly diagnosed FLT3-ITD positive and NPM1 wild-type AML pediatric patients.

This study is a linked trial to the CHIP-AML22/Master protocol. Patients will start in the CHIP-AML22/Master study and if they are FLT3-ITD positive and NPM1 wild-type, can be enrolled in the CHIP-AML22/Quizartinib study.

ELIGIBILITY:
Inclusion criteria:

1. Enrollment on CHIP-AML22/Master:

   Patients must be enrolled on the CHIP-AML22/Master prior to enrollment on CHIP-AML/Quizartinib linked-trial, and may have received a diagnostic work-up according to the master protocol. Induction treatment can be started as standard of care.
2. FLT3-ITD+ and wild-type NPM1:

   Presence of FLT3-ITD+ and NPM1 wild type in bone marrow or peripheral blood provided by the local laboratories, as part of standard of care diagnostics. The results of FLT3-ITD testing must be obtained prior to the first dose of quizartinib (e.g., Induction course 1, Day 10).
3. Age:

   Patients must be from 1 month to ≤ 18 years old at initial diagnosis
4. Performance status Karnofsky performance status score of >50% for subjects >16 years of age, and a Lansky performance status score of >50% for subjects ≤16 years of age.
5. Organ function criteria:

   These criteria must be met based on the results before start of any chemotherapy (e.g., MEC) a. Adequate Renal Function Defined as:

   • Calculated eGFR ≥ 50 mL/min/1.73 m2 using the Schwartz formula. b. Adequate Liver Function Defined as:
   * Total or direct (conjugated) bilirubin < 1.5xULN for age (≤ 5xULN if related to leukemic involvement), AND
   * Aspartate transaminase (AST) and alanine transaminase (ALT) <5xULN (<10×ULN if related to leukemic involvement)
6. Life expectancy: > 6 weeks
7. Pregnancy test:

   Serum/urine pregnancy test (for all girls ≥ age of menarche) negative within 2 weeks prior to enrollment on the quizartinib linked-trial.
8. Taking quizartinib:

   Patients must be able to reliably swallow or administer quizartinib by NG tube.
9. Informed consent:

   Written informed consent/assent for the quizartinib linked trial from patients and/or from parents or legal guardians for minor patients, according to local law and regulations.

   General exclusion criteria:
   1. Patients with only extramedullary disease
   2. Uncontrolled or significant cardiovascular disease, including -Diagnosed or suspected congenital long QT syndrome

      -History of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes); any history of arrhythmia will be discussed with sponsor, the national coordinator and C.I.the prior to subject's entry into the study.

      -QT interval corrected >450 ms: QTc interval corrected with Fridericia's formula (QTcF) for subjects ≥ 6 years of age at the time of enrollment.

      -Left ventricular systolic dysfunction (LVSD), defined as ejection fraction (EF) below 55% during the screening for the CHIP-AML22/Master protocol.

      -History of uncontrolled angina pectoris or myocardial infarction within 6 months.

      -History of second (Mobitz II) or third degree heart block (subjects with pacemakers are eligible if they have nohistory of fainting or clinically relevant arrhythmias while using the pacemaker).

      -Heart rate <50 beats/minute on ECG during the screening for the CHIP-AML22/Master protocol (In case,adolescents with a normal sinusoidal rhythm and no evidence of other cardiac dysfunction will be discussed with sponsor, the national coordinator and C.I. the prior to subject's entry into the study.)

      -Uncontrolled hypertension (e.g., systolic blood pressure and /or diastolic blood pressure that is, on repeated measurement, at or above the 95th percentile for sex, age, and height).
      * History of complete left bundle branch block.
      * History of New York Heart Association Class 3 or 4 heart failure.
   3. Known history of HIV or active clinically relevant liver disease (e.g., active hepatitis B or active hepatitis C)
   4. Underlying GI disease that may affect absorption of study drug
   5. Use of strong or moderate CYP3A inducers will be prohibited throughout the duration of the study. Strong CYP3A4 inhibitors will be allowed with a concomitant dose reduction of quizartinib with the exception during the safety run-in.
   6. History of hypersensitivity to any of the study medications or their excipients.
   7. Other serious illnesses or medical conditions, that will likely make it impossible to complete treatment according to protocol (e.g., patients who should not be given any of the study medications based on the SmPC)
   8. Currently participating in other investigational interventional procedures, if it interferes with any endpoints of the quizartinib trial.

2) Additional exclusion criteria during safety run-in:

1. Patients with CNS3 disease
2. Using strong CYP3A4 inhibitors (If patient can stop using strong CYP3A4 inhibitors, he/she will be allowed to enroll. In such case, no washout is required for the strong CYP3A4 inhibitor)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2032-06 (Estimated)

PRIMARY OUTCOMES:
Primary objective (efficacy) | 2 induction courses (maximum of 56+/-2 days per course)
  The percentage of patients with (Minimal Residual Disease) MRD levels <0.1% (MRD negativity) after up to 2 courses of induction chemotherapy plus quizartinib, as measured in the bone marrow using multiparameter flow cytometry (MFCM) before start of consolidation therapy, in the evaluable population for response.
  o Patients to be evaluated at baseline, end of cycle 1, and end of cycle 2
Primary objective (safety) | 2 induction courses (maximum of 56+/-2 days per course)
  Incidence of Dose-Limiting Toxicities (DLTs) assessed during Induction course 1 and 2 (until day 56 of each course) for the DLTs evaluable patients.

SECONDARY OUTCOMES:
Secondary objectives (efficacy_1) | 2 induction courses (maximum of 56+/-2 days per course)
  Morphological overall response rate (ORR)
Secondary objectives (efficacy_2) | Multiple time points, last time point after continuation treatment (1.5 years)
  MRD by multiparameter flow cytometry (MFCM)
Secondary objectives (efficacy_3) | 3 years
  Event free survival (EFS)
Secondary objectives (efficacy_4) | 3 years
  Overall survival (OS)
Secondary objectives (efficacy_5) | 3 years
  Disease free survival (DFS)
Secondary objectives (efficacy_6) | 3 years
  Duration of response
Secondary objectives (efficacy_7) | 3 years
  Cumulative incidence of relapse (CIR)
Secondary objectives (efficacy_8) | 1 year
  Number and percentage of patients actually being treated with hematopoietic stem cell transplantation (HSCT)
Secondary objectives (efficacy_9) | 1.5 years
  Number of patients starting and completing continuation treatment post-HSCT.
Secondary objectives (safety) - Adverse Events, Laboratory Abnormalities and cumulative incidence of non-relapse mortality | 1.5 years
  Safety and tolerability of combining quizartinib with conventional treatment and quizartinib given as single-agent after HSCT.
  * Adverse events (AEs), as characterized by type, frequency, severity (as graded using CTCAE, v5.0).
  * Laboratory abnormalities (including time to recovery of ANC and PLT), electrocardiograms and changes in vital signs as characterized by type, frequency, severity and timing will be tabulated, and reported as AEs when considered clinically significant by the investigator.
  * The cumulative incidence of non-relapse mortality, defined as the cumulative probability of non-relapse mortality, with time calculated between start of study treatment and death due to other causes than relapsed or refractory leukemia, accounting for competing events.
Pharmacokinetics (PK_1) | 1.5 years
  Population PK analysis to estimate AUC (tau) for quizartinib and AC886
Pharmacokinetics (PK_2) | 1.5 years
  Population PK analysis to estimate Cmax for quizartinib and AC886
Pharmacokinetics (PK_3) | 1.5 years
  Population PK analysis to estimate clearance (CL/F) for quizartinib.
Pharmacokinetics (PK_4) | 1.5 years
  Population PK analysis to estimate volume of distribution (Vss/F) for quizartinib.
Palatability of quizartinib formulations | 1.5 years
  Patients and/or parents or legal guardians will answer using a Hedonic scale for the taste and ability to swallow the medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Gertjan Kaspers, Prof. Dr., Study Chair — Pediatric Oncologist; Michel Zwaan, Prof. Dr., Study Director — Head Trial and Data Center
Locations (1):
- Princess Máxima Center for pediatric oncology, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data will be used to generate a publication
Supporting Information: CSR
Time Frame: Primary CSRs may be completed earlier when the primary objective is completed and may be followed by a final CSR not later than 6 months after the LPLV.
Access Criteria: A summary of the study results will be made public via clinicaltrials.gov as well as to Ethical committees/ Health Authorities and all participating patients by providing them through their treating physicians a patient letter with a summary of the results.